CLINICAL TRIAL: NCT06414915
Title: A Single-arm, Open, Single-center, Prospective and Exploratory Clinical Study of Surufatinib Combined With Tislelizumab in the Treatment of Advanced Lung Cancer With Neuroendocrine Differentiation
Brief Title: Surufatinib Combined With Tislelizumab in Advanced Lung Cancer With Neuroendocrine Differentiation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Puyuan Xing, Chief Medical Officer, National Cancer Center, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-NEN110
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: NSCLC
Keywords: NSCLC; neuroendocrine differentiation; Surufatinib; Tislelizumab
MeSH Terms: interventions — surufatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib + tislelizumab (Experimental)
  Interventions: Drug: Surufatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Surufatinib — 250 mg, po, qd, q3w
Drug: Tislelizumab — 200mg, iv, q3w

SUMMARY:
Currently, there are no standard treatment and relevant exploration for NSCLC patients with NED. The study aims to explore the efficacy and safety of surufatinib combined with tislelizumab in the treatment of NSCLC with NED, in order to provide a new treatment option for NSCLC patients with NED.

DETAILED DESCRIPTION:
This is a single-arm, open, single-center, prospective and exploratory clinical study. We planned to enroll 29 patients who would receive surufatinib plus tislelizumab until disease progression, intolerance, or withdrawal of consent. The study aims to explore the efficacy and safety of surufatinib combined with tislelizumab in the treatment of NSCLC with NED, in order to provide a new treatment option for NSCLC patients with NED.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed locally advanced or metastatic unresectable lung cancer (IIIB-IV) with an abnormal NED or NE phenotype (without neuroendocrine morphologic features and positive immunohistochemical expression of at least one neuroendocrine marker (CD56, CgA, Syn));
* Have at least one measurable lesion according to RECIST v1.1;
* ECOG performance status: 0-1;
* Patients who were deemed by the investigator to be eligible for first-line single-agent immunotherapy or who progressed on first-line standard therapy;
* Urine protein < ++ . If Urine protein ≥ ++ ,the amount of urine protein in 24 hours ≤1.0g;
* Expected survival time > 3 months;

Exclusion Criteria:

* Pulmonary neuroendocrine tumors (typical carcinoid, atypical carcinoid, small cell carcinoma, large cell neuroendocrine carcinoma);
* Prior anti-VEGF/VEGFR-targeted therapy or anti-PD (L)1 antibody;
* Have uncontrolled hypertension, defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mm Hg, while under anti-hypertension treatment;
* Patients with active ulcer, intestinal perforation and intestinal obstruction;
* With active bleeding or bleeding tendency;
* Severe history of cardiovascular and cerebrovascular diseases;
* Other malignancies diagnosed within the previous 5 years, except basal cell carcinoma or cervical carcinoma in situ after radical resection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | approximately 1 years
  time from first-dose to the first documented disease progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | approximately 1 years
  the proportion of patients with complete response or partial response, using RESIST v1.1
Disease Control Rate (DCR) | approximately 1 years
  the proportion of patients with complete response, partial response or stable disease, using RESIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Puyuan Xing, Doctorate, Principal Investigator — Department of Medical Oncology, National Cancer Center, China

IPD SHARING:
Plan to Share IPD: No